CLINICAL TRIAL: NCT05468593
Title: Patient Reported Outcomes After Hepatic Artery Infusion Pump Placement
Brief Title: Patient Outcomes After Hepatic Artery Infusion Pump Placement
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cornelius A. Thiels, Principal Investigator, Mayo Clinic
Other Study IDs: 22-003190
Record Dates: First submitted 2022-07-12; First posted 2022-07-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Liver Metastases; Colorectal Cancer
Keywords: Hepatic Artery Infusion; Pump; Hepatic Artery Infusion Chemotherapy; Unresectable Colorectal Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the surgical outcomes and the quality of life (QOL) in patients undergoing hepatic artery infusion pump placement for colorectal liver metastases (CRLM).

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive a Hepatic Artery Infusion Pump at Mayo Clinic Rochester for liver metastases from colorectal cancer.
* Written consent.

Exclusion Criteria:

* Absence of written consent.
* Systemic disease.
* Pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal liver metastases (CRLM) being offered Hepatic Artery Infusion Pump placement and subsequent Hepatic Artery Infusion Chemotherapy at Mayo Clinic Rochester will be evaluated to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Baseline prior to surgery.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 2.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 7.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 14.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 30.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 60.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 90.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 120.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 150.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.
Quality of Life | Postoperative day 180.
  Self-reported quality of life and recovery from surgery using a questionnaire to investigate changes over time.

SECONDARY OUTCOMES:
Time to start chemotherapy | 1 month postoperatively
  Number of days following hepatic artery infusion pump placement until chemotherapy is started
Surgical outcomes | 1 month postoperatively
  Complications with hepatic artery infusion pump placement
Surgical outcomes | 6 month postoperatively
  Complications with hepatic artery infusion chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Thiels, DO, MBA, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials